CLINICAL TRIAL: NCT03980431
Title: Safety and Clinical Value of 18Fluorine-labeled Boron Tyrosine PET/CT in Patients With Brain Tumors
Brief Title: FBY PET/CT in Patients With Brain Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-FBY PET/CT
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; FBY-Positron Emission Computed Tomography (FBY-PET); glioma; brain metastasis
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Intervention Model Description: A single dose of 0.10 mCi/kg FBY will be intravenously injected and PET examination will carry out 30 minutes later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBY in suspected malignant brain tumor (Experimental): This arm investigates the metabolic characteristics of FBY in suspected malignant brain tumor patients who consider for surgical operations. A single dose of 0.10 mCi/kg FBY will be intravenously injected and PET examination will carry out 30 minutes later. Surgical operations, if recommended after multiple examination, will be carried out within 1 week after FBY PET scan.
  Interventions: Diagnostic Test: FBY PET Examination
- FBY in suspected recurrent glioma (Experimental): This arm investigates the value of FBY to differentiate tumor progression from pseudoprogression. A single dose of 0.10 mCi/kg FBY will be intravenously injected and PET examination will carry out 30 minutes later. Surgical operation, MRI follow up or change of treatment strategy, according to specific conditions, will be recommended for the definitive diagnosis as well as the management of patients.
  Interventions: Diagnostic Test: FBY PET Examination

INTERVENTIONS:
Diagnostic Test: FBY PET Examination — A single dose of 0.10 mCi/kg FBY will be intravenously injected and PET examination will carry out 30 minutes later.

SUMMARY:
This study is an open-labeled phase II diagnostic clinical trial to explore the safety and clinical value of FBY in suspected adult brain tumor patients. The investigation regarding the clinical value of FBY includes 1) the metabolic characteristics of FBY in suspected malignant brain tumors; 2) role of FBY to differentiate tumor progression from pseudoprogression. A single dose of 0.10 mCi/kg FBY will be intravenously injected for PET examination. Quantitative features will be extracted to analysis the PET images. Cranial MRI (with contrast enhancement) will also performed as diagnostic comparison with FBY. For patient who took surgery after multiple examination, histopathology, molecular pathology and LAT-1 immunohistochemistry will also be obtained.

DETAILED DESCRIPTION:
FBY is a new PET tracer derived from tyrosine, with the carboxyl group replaced by boron trifluoride, and is transferred across cell membrane through LAT-1. LAT-1 is a sodium independent amino acid transporter and is highly expressed in tumor cells. Considering the significant role in cancer development as well as in nutrient delivery, FBY could be a promising PET tracer to reflect altered metabolism in tumors.

This study aim to observe the safety of FBY, and investigate the diagnostic value of FBY in the patient with suspected brain tumors. Patients who meet the eligibility criteria are included in clinical trials after fully communicating the condition, explaining the benefits and risks of clinical trials, clarifying the patient's willingness to include the clinical trial, and signing informed consent. The cohort number, FBY administrative dose, imaging protocols are decided based on the investigators' preliminary data. The diagnosis and post-examination treatment are based on the recommended guideline, combined with the subject's own situation for standardized diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have suspected diagnosis of brain tumors, based on clinical performance and MRI results.
* 2. Meet the indications for PET examination, show a clear indication and no contraindications;
* 3. Have a performance status of score ≥70 on KPS scale or score 0-1 points on ECOG scale, a relatively good general situation;
* 4 Does not appear agonal stage, deep coma, over grade 2 major organ dysfunction (heart, lung, liver, kidney and other major organ include), acute or life-threatening status of infection;
* 5. Be ≥ 18 years of age on day of signing informed consent.
* 6. Be willing and able to understand the research content and provide written informed consent/assent for the trial.

Exclusion Criteria:

* 1. Have a history of imaging agent allergies;
* 2. Does not meet the PET-CT scan sedation requirements, or there are contraindications for PET-CT examination;
* 3. Be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial;
* 4. Unable to adhere strictly to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
standardized uptake value (SUV) for FBY | 1 week.
  SUV reflects the uptake of PET tracers, and quantitative imaging features such as SUVmax, SUVmean, and visually-assessed features will be measured in the evaluation of tumors.

SECONDARY OUTCOMES:
Adverse events | 1 week.
  Adverse event within 1 week after FBY injection will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenbin Ma, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 Brain and Other CNS Cancer Collaborators. Global, regional, and national burden of brain and other CNS cancer, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Apr;18(4):376-393. doi: 10.1016/S1474-4422(18)30468-X. Epub 2019 Feb 21. PMID 30797715
- [Background] Rohrich M, Huang K, Schrimpf D, Albert NL, Hielscher T, von Deimling A, Schuller U, Dimitrakopoulou-Strauss A, Haberkorn U. Integrated analysis of dynamic FET PET/CT parameters, histology, and methylation profiling of 44 gliomas. Eur J Nucl Med Mol Imaging. 2018 Jul;45(9):1573-1584. doi: 10.1007/s00259-018-4009-0. Epub 2018 May 7. PMID 29732524
- [Background] Chansaenpak K, Wang M, Wang H, et al. Preparation of [18F]-NHC-BF3 conjugates and their applications in PET imaging. RSC Advances, 2017, 7(29): 17748-17751.
- [Derived] Li Z, Kong Z, Chen J, Li J, Li N, Yang Z, Wang Y, Liu Z. 18F-Boramino acid PET/CT in healthy volunteers and glioma patients. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3113-3121. doi: 10.1007/s00259-021-05212-7. Epub 2021 Feb 15. PMID 33590273